CLINICAL TRIAL: NCT05096078
Title: The Effect of Circuit Exercise Program on Cognitive Function, Functional Exercise Capacity, Mobility, Depression and Quality of Life in Women With Gestational Diabetes
Brief Title: The Effect of Circuit Exercise Program in Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Miray Budak, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GestationalDM.Exer.Cog.
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Circuit Exercise; Cognition
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Group (Active Comparator): Individuals will receive only dietary treatment that the dietitian deems appropriate for 6 weeks.
  Interventions: Other: Diet
- Exercise Group (Experimental): In addition to the 6-week diet program that the dietitian deems appropriate, a circuit exercise program will be applied for 6 weeks. The circuit exercise program will consist of a medium-intensity circuit training for 50 minutes, 3 days a week, detailing the main muscle groups of the patients (chest, back, biceps, triceps, deltoid, quadriceps, thigh and calf muscles). Exercise intensity will be monitored using Borg's scale of perceived exertion, with a target intensity of 12 to 14. 8 exercises will be given in a continuous, circuit-type manner with short 1-minute rests.
  Interventions: Other: Diet; Other: Exercise

INTERVENTIONS:
Other: Diet — Special diet program for gestational diabetes
Other: Exercise — The circuit exercise program will consist of a medium-intensity circuit training for 50 minutes, 3 days a week, detailing the main muscle groups of the patients (chest, back, biceps, triceps, deltoid, quadriceps, thigh and calf muscles). Exercise intensity will be monitored using Borg's scale of perceived exertion, with a target intensity of 12 to 14. 8 exercises will be given in a continuous, circuit-type manner with short 1-minute rests.
  Arms: Exercise Group

SUMMARY:
Gestational diabetes (GDM) is defined as 'pregnancy-onset or first noticed glucose intolerance'. The aim of this study is to investigate the effect of circuit exercise program applied in addition to diet therapy on cognitive function, functional exercise capacity, mobility, depression and quality of life in women with gestational diabetes. 60 female participants between the ages of 18-35 who meet the inclusion criteria will be included in the study. Participants will be randomly divided into 2 groups as diet group (n=30) and exercise group (n=30). All participants will receive GDM-specific dietary therapy for 6 weeks. In addition to diet therapy, individuals in the exercise group will be given a circuit exercise program for 6 weeks. Participants will be evaluated for blood values, cognitive status and functionality at the baseline and 6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with gestational DM
* being between the ages of 18-35
* being in 24-32 weeks of pregnancy
* being inactive physical activity level - (<300 MET weeks/day)

Exclusion Criteria:

* Diagnosed with diabetes before pregnancy
* have given birth before
* Multiple Pregnancy (>2)
* Intrauterine growth restriction
* Preeclampsia
* having high risk of preterm labor and on strict bed rest
* treatment with insulin or oral hypoglycemic agents during pregnancy
* Other significant severe or poorly controlled medical conditions (thyroid disease, cardio-respiratory disorders, ...)
* taking medications that affect cognitive function, including corticosteroids, anti-depressants, or anti-epileptics

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Blood count test 1 | 6 weeks after baseline
  Fasting blood glucose (FBG) value will be recorded.
Blood count test 2 | 6 weeks after baseline
  Postprandial blood glucose (PBG) value will be recorded.
Blood count test 3 | 6 weeks after baseline
  HbA1c value will be recorded.
Blood count test 4 | 6 weeks after baseline
  Total cholesterol (T-col) value will be recorded.
Blood count test 5 | 6 weeks after baseline
  High-density lipoprotein cholesterol (HDL) value will be recorded.
Blood count test 6 | 6 weeks after baseline
  Low-density lipoprotein cholesterol (LDL) value will be recorded.
Blood count test 7 | 6 weeks after baseline
  Insulin value will be recorded.
Blood count test 8 | 6 weeks after baseline
  Triglyceride (TG) value will be recorded.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale | 6 weeks after baseline
  It is a screening scale developed to evaluate the early stages of cognitive impairment. Min score is 0, max score is 30. High scores mean a better outcome.
WMS Number Range Test | 6 weeks after baseline
  In the forward number range, the patient is asked to repeat the numbers told to her in the same order, and in the backward number range, the patient is asked to repeat the said numbers from the end to the beginning. High scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, PhD, Study Director — Medipol University; Saadet Turhan, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)